CLINICAL TRIAL: NCT03369353
Title: Precision Diagnostics in Inflammatory Bowel Disease, Cellular Therapy and Transplantation (The PREDICT Trial)
Acronym: PREDICT
Status: Enrolling by invitation | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Leslie Kean, MD, PhD, Boston Children's Hospital
Other Study IDs: P00030890
Record Dates: First submitted 2017-09-26; First posted 2017-12-12 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Graft Vs Host Disease; Inflammatory Bowel Diseases; Functional Gastrointestinal Disorders
Keywords: Bone Marrow Transplantation; Graft Vs Host Disease; Inflammatory Bowel Diseases; Functional Gastrointestinal Disorders; Cellular Therapy
MeSH Terms: conditions — Graft vs Host Disease; Inflammatory Bowel Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Stool Biopsy tissue from endoscopy Cerebrospinal Fluid Bone marrow aspirate Tissue samples from clinical biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the Precision Diagnosis in Inflammatory Bowel Disease, Cellular Therapies, and Transplantation (PREDICT) trial is to apply a systems-biology approach to enable precision diagnostics for the key immunologic outcomes for patients with Inflammatory Bowel Disease, Cellular Therapeutics and Transplantation. This approach will deepen the understanding of the molecular mechanisms driving auto- and allo-immune diseases and serve as a critical platform upon which to design evidence-based treatment paradigms for these patients.

This research study will examine the immunology of auto- and allo-immune gastrointestinal disturbances such as Inflammatory Bowel Disease (IBD), Graft-versus-Host Disease (GVHD), and Functional Gastrointestinal Disorder (FGID), as well as the immune manifestations after CAR-T and other cellular therapeutics. The Investigators seek to use blood and tissue samples in order to better understand the mechanisms driving these diseases and their therapies.

The Investigators further hypothesize that longitudinal systems-based immunologic analysis will enable the patient-specific determination of the molecular evolution of IBD, GVHD and the response to cellular therapeutics, as well post-transplant defects in protective immunity, and determine which pathways, when perturbed, can cause clinical disease. The discovery of these pathways will lead to improved diagnostic, prognostic and treatment approaches, and to personalized therapeutic decision-making for these patients.

DETAILED DESCRIPTION:
Hypotheses:

Hypothesis #1: The Investigators hypothesize that they can define the molecular mechanisms responsible for Inflammatory Bowel Disease (IBD) and gastrointestinal (GI) acute GVHD and differentiate it from other inflammatory disorders by using advanced immunologic analysis including flow cytometry, TCR deep sequencing and transcriptomics.

Hypothesis #2: The Investigators further hypothesize that longitudinal systems-based immunologic analysis will enable the patient-specific determination of the molecular evolution of IBD as well as acute and chronic GVHD as well post-transplant defects in protective immunity, and determine which pathways, when perturbed, can cause clinical disease. The discovery of these pathways will lead to improved diagnostic, prognostic and treatment approaches, and to personalized therapeutic decision-making for patients undergoing hematopoietic stem cell transplantation (HCT).

Hypothesis #3: We hypothesize that we can define the molecular mechanisms, phenotypic and functional immunologic characteristics involved in distinct determinants of adoptive cellular therapies, including the efficacy, longevity and toxicity associated with cellular therapy. Longitudinal characterization of cellular therapeutics and the endogenous immune response they elicit using advanced immunologic analysis including flow cytometry, mass spectrometry, TCR deep sequencing and single-cell transcriptomics will allow identification and distinction of pathways critical for efficacy and toxicity and enable subsequent therapeutic modulation.

Hypothesis #4: We hypothesize that differences in the gut microbiome of patients with IBD and recipients of HCT play a major role in disease severity and overall clinical outcomes in both diseases (e.g. bacteremia, unexplained fevers, mortality). The longitudinal characterization of the gut microbial communities by next generation sequencing will allow for detection of sequential microbial changes that coincide with observed clinical changes. the discovery of significant changes in the microbiome that are repeatedly observed with a particular clinical outcome will lead to better mechanistic understanding of its pathophysiology and inform future diagnostic and preventive approaches.

Hypothesis #5: We hypothesize that immune dysregulation associated with a wide range of disorders will alter the immune response to vaccines, compounding susceptibility to infectious diseases in these populations. Specifically, HCT and solid organ transplant recipients, as well as patients with active or recent history of malignancy, or autoimmune diseases may have reduced T and B cell responses to SARS-CoV-2 vaccination due to the effect of disease pathophysiology or treatment regimens on immune function. Comprehensive serologic analysis, high parameter flow cytometry, and T and B cell RNA sequencing will enable longitudinal analysis of neutralizing antibody titers and antigen-specific T and B cell expansion, phenotype, diversity, and survival following vaccination in these patient populations, as well as in related and unrelated healthy controls. These data will provide mechanistic insight into how immune impairment in these disorders contributes to poor responses to infections. as SARS-CoV-2 is a pathogen to which much of the population remains naïve, this represents a unique opportunity to study the immune response to a novel challenge in immunocompromised individuals. Moreover, these findings will inform public health guidelines on how to improve measures to protect vulnerable populations from preventable disease.

Aims:

Specific Aim #1: To identify the mechanisms specific for IBD and GI acute GVHD and delineate it from other inflammatory disorders.

Objective 1: Perform flow cytometry, TCR deep sequencing and whole transcriptome analysis on T cells purified from GI tissue samples taken from patients who undergo endoscopy for presumed GI GVHD, inflammatory bowel disease (IBD), and functional gastrointestinal disease (FGID).

Objective 2: Perform flow cytometry, TCR deep sequencing and transcriptome analysis on T cells from the peripheral blood at the time of endoscopy in patients diagnosed with GI GVHD, IBD, and FGID.

Specific Aim #2: Characterize the immunologic dysregulation responsible for IBD, acute GVHD, chronic GVHD and defects in protective immunity in patients undergoing HCT.

Objective 1: Perform longitudinal immune analysis on T cells and B cells purified from patients with IBD and those undergoing allogeneic HCT. For transplant patients, we will compare T and B cell immunity in patients who develop acute and chronic GVHD, relapse, and infectious complications post-transplant and compare to patients without these complications.

Objective 2: Perform microbiome analysis longitudinally in patients with IBD and those undergoing HCT to determine the impact of microbiome alterations in the development of post-transplant complications.

Specific Aim #3: Identify the molecular and cellular immunologic mechanisms involved in determining the clinical response to cellular therapies and distinguish pathways critical to a successful anti-tumor response from those involved in adverse effects.

Objective 1: Characterize the cellular product prior to administration and track its distribution, kinetics, persistence and function longitudinally in vivo in the patient's peripheral blood and when applicable bone marrow, CSF and other tissues, using qPCR-based transgene detection (if applicable), flow cytometry, mass cytometry, TCR deep sequencing and whole transcriptome analysis on T cells and other immune cells contained in the cellular product.

Objective 2: Longitudinally interrogate the interplay of the cellular therapy with the endogenous immune system and delineate the role of the endogenous immune response in the efficacy, persistence and toxicity of cellular therapy, using flow cytometry, mass cytometry, TCR deep sequencing, whole transcriptome analysis on endogenous immune cells and analysis of soluble factors and antibodies.

Specific Aim #4:Characterize the antigen-specific adaptive immune response to SARS-CoV-2 vaccination in patients with immune dysregulation due to cancer, transplantation, or autoimmune disease and identify mechanisms underlying impaired generation of durable immunity.

Objective 1: Perform comprehensive longitudinal analysis of serologic immunity pre- and post-vaccination, including to booster vaccines, in patients and healthy controls, including assessment of SARS-CoV-2 specific antibody levels and neutralizing antibody titers.

Objective 2: Use high parameter flow cytometry, single cell RNA sequencing (scRNAseq), and T and B cell repertoire analysis to characterize the longitudinal development of antigen-specific T and B cell memory to SARS-CoV-2 following vaccination and subsequent booster vaccines in patients and healthy controls.

Objective 3: Assess the ability of sera and cloned antibodies from patients to respond to bind and neutralize viral variants, as compared to that of healthy controls.

Background and Significance:

IBD: Inflammatory bowel disease (IBD) which includes Crohn's Disease (CD) and Ulcerative Colitis (UC), is a chronic complex gastrointestinal (GI) autoimmune condition that inflicts 1.4 million people in the united states1. The incidence and prevalence of both CD and UC are increasing over time and encompassing larger areas of the world1,2. In addition, pediatric IBD comprises 25% of all diagnosed IBD, relegating the child to a lifetime of gastrointestinal disease and exposure to immunosuppression especially during a period meant for growth and development. Despite ongoing research into the pathogenesis and genetic abnormalities, the mechanism behind IBD development and progression is not well understood. Standard therapies still rely on steroids, other non-specific immunosuppression (such as methotrexate and azathioprine), and anti-TNF biologics. Although newer therapies such as agents that block cytokines and leukocyte trafficking are emerging, no universally successful treatments have been identified. Thus, relapsing forms of IBD continue to lead to systemic compromise in nutritional absorptive capacity, anemia, and often, to the need for surgical interventions. Deciphering the mechanisms driving the unique subtypes of IBD (even within UC and CD) then optimizing treatment based on the underlying systemic dysregulation is a critical unmet need in the field. While the underlying immune mechanism of IBD remains undetermined, there is significant data to suggest that IBD may represent an inappropriate immune response towards self antigens and commensal microbiota in a genetically susceptible host3. Thus, murine colitis models suggest that mucosal inflammation results from pathologic T helper- (Th) cell responses, along with regulatory cell defects. These data have emerged from experiments in IL-2 deficient mice4, IL-10 deficient mice5, TGF-beta6, and TGF-betaGRII dominant negative transgenic mice7. The pathogenesis also includes an exaggeration in effector cell responses, which have emerged from experiments in Stat4 transgenic mice8 and TNFARE mutant mice9. More recently human cytokine analysis suggests that despite clinical similarities, each subtype of IBD show distinctive cytokine profiles10. Although initial studies have begun to target specific effector T cell pathways11, the application of target organ transcriptomics is in its infancy and individual targetable pathways are still elusive.

HCT: Allogeneic HCT is an effective treatment for patients with malignant and non-malignant hematologic diseases. However, this treatment is complicated with high rates of morbidity and mortality limiting its broader application. The leading causes of post-transplant morbidity and mortality include acute and chronic GVHD, relapse and infectious disease. The goal of the PREDICT trial is to apply a systems approach to understanding the mechanisms driving these complications, such that evidence-based treatment strategies can be devised.

Acute GVHD: Acute GVHD is mediated by donor-derived allo-reactive T cells becoming activated and resulting in cytotoxicity against host cells12,13 as well as cytokine-mediated tissue damage. Moderate to severe acute GVHD can occur in up to 60% of patients undergoing HCT and the more severe forms have been associated with mortality rates >50%14-17. The most common sites of the immune-mediated tissue damage are the liver, skin, and gastrointestinal (GI) tract. GI GVHD occurs in 40-50% of HCT patients and is the major cause of morbidity and mortality from this disease17.

The diagnosis of GI GVHD is derived from clinical and histopathological findings. GVHD can occur in both the upper and lower GI tract leading to symptoms of diarrhea, abdominal pain, nausea, vomiting, and/or anorexia12. Histopathological diagnostic criteria for GI GVHD includes identification of crypt cell apoptosis, crypt destruction and/or mucosa denudation18. Unfortunately, the severity of GVHD on histology is poorly correlated with the clinical course of the disease.

While GI GVHD is a common complication following HCT there remain many barriers to its consistent and accurate diagnosis. First, diagnosis is dependent on appropriate tissue sampling. Visible lesions are frequently absent19 and endoscopic findings can be diffuse and nonspecific. There is also no consensus on the optimal location of the GI tract for biopsies or number of biopsies needed to secure a diagnosis. There is also frequent discordance between biopsy specimens from the upper and lower GI tract20. Second, patients presenting early in the course of GVHD may have subtle histopathological findings that may be missed or not yet present. At the onset of GVHD few apoptotic cells may be seen and crypt loss and mucosal damage may yet to have occured18. Lastly, there are also confounding factors that can lead to the misdiagnosis of GVHD that include conditioning regimen related toxicity, concomitant infections, and medications which can all cause focal inflammation of the GI tract. In the first 20 days following a myeloablative conditioning regimen diffuse apoptosis can be seen mimicking acute GVHD21. Clostridium difficile and cytomegalovirus infections can also have similar clinical and histopathological presentations22. Use of mycophenolate mofetil23 and proton pump inhibitors24 have also been found associated with GI tract apoptosis that can be misdiagnosed as GVHD. All of these factors lead to the high degree of inter-observer variability in the histological diagnosis of GVHD18,25 and poor correlation with the clinical observations, illustrating the need for more sensitive and specific methods of diagnosis.

There have been recent advances in the identification of biomarkers in GVHD that have diagnostic and prognostic significance. IL-8, IL-2 receptor-alpha, tumor necrosis factor receptor-1 (TNF-1), hepatocyte growth factor (HGF), elafin, regenerating islet-derived 3-alpha (reg-3alpha), TIM3, IL-6, ST2, B-cell activating factor (BAFF), IL-33, CXCL10, and CXCL11 have all been found to have utility in predicting the development of GVHD26-28. While these biomarkers have been identified they have not been extensively validated and are yet to be clinically adopted as a guide to alter treatment. Moreover, the biomarkers discovered thus far are often the result of downstream pathway perturbations and discovering the upstream dysregulation that occurs earlier in the course of the disease may be valuable in developing diagnostic or prognostic models that could lead to trials aimed at altering the natural course of the disease.

Our group has previously shown that by using advanced immunologic analysis including flow cytometry, and whole transcriptome analysis, we can identify previously unrecognized molecular pathways active in GVHD29-31. We anticipate that by utilizing a systems immunology approach in patients with acute GVHD we will be able to identify pathways that have diagnostic and prognostic value. This may enhance our diagnostic capacity and most importantly, allow us to individualize management of patients based on their specific immunologic profiles.

Chronic GVHD: CGVHD occurs in 40-60% of transplant patients32-35 with the incidence of this disease rising in the past 2 decades36 chronic GVHD causes significant mortality, and in those patients that survive, it can result in profound effects on quality of life37-40. Despite the increased frequency of chronic GVHD, accurate diagnosis and evidence-based therapy is still lacking. Thus, while chronic GVHD biomarkers have been identified there have yet to be any that qualify for clinical application41. Moreover, these biomarkers often represent end-stage pathway perturbations and may result from nonspecific inflammation and tissue damage as well as counter-regulatory mechanisms. In addition to the challenges in diagnosis, there are significant treatment challenges as well: Thus, treatment of chronic GVHD has not changed significantly over the past few decades. First line therapy remains corticosteroids with or without calcineurin inhibitiors (CNIs)42-44 and unfortunately, approximately 50% of patients will fail and require second line treatment45,46 with failure-free survival at 2 years following second-line therapy being only 25%47. These data underscore the significant unmet needs in this field, both for molecular diagnostics and evidence-based treatment paradigms.

Protective Immunity: In addition to the challenges of acute and chronic GVHD, patients undergoing HCT and those with IBD face other toxicities as well, many of which are related to dysfunctional immune reconstitution after transplant. However, although the phenomenology of the many defects in protective immunity (both against infectious pathogens and against leukemia relapse) is well-documented, the causative molecular mechanisms remain unknown. To address these questions, our group and others have begun to perform detailed assessments of immunologic reconstitution after HCT including the application of new T Cell Receptor (TCR) and B cell Receptor (BCR) deep-sequencing technologies30,48-54. These technologies allow the investigation of the breadth and depth of post-transplant immune reconstitution at a level of molecular detail not previously possible and hold the promise of deepening our understanding of the impact of infectious pathogens on global immune health and immune reconstitution. The widespread application of these technologies, and their intersection with detailed assessment of immune phenotype and function can provide novel insights about the state of immune health in transplant patients, and holds the promise of identifying patients in need of novel interventions to improve their post-transplant immune reconstitution.

The goal of the PREDICT trial is to apply a systems-biology approach to enable precision diagnostics for the key immunologic outcomes post-transplant. This approach will deepen our understanding of the molecular mechanisms driving the most deadly post-transplant complications, and serve as a critical platform upon which to design evidence-based treatment paradigms for transplant patients.

Cellular Therapy: Novel adoptive cell therapies are increasingly entering clinical trials and are available as FDA approved biologics, thereby providing a therapeutic option for previously refractory patients. This broad and exciting field includes chimeric-antigen receptor (CAR) T cells directed against a variety of antigens55, T cells genetically modified to express TCRs56,57, cytokine-stimulated NK-cells58, as well as tumor vaccine approaches with endogenous, irradiated tumor samples59 or immune cells pulsed with tumor antigen.60 Chimeric antigen-receptor T cells have led to dramatic responses, particularly in patients with CD19+ B-cell malignancies61-64, leading to FDA approval of several products. While unprecedented clinical remissions can be achieved initially, the approach is frequently limited by the durability of the response and CAR T cell persistence with an EFS of 50% at 12 months after infusion61, tumor escape mechanisms65 and significant toxicity involving cytokine release syndrome, neurologic toxicity66. In the context of CAR T cell therapy, key factors for successful application have been identified and include incorporation of a costimulatory signaling mechanism67,68, association of in vivo CAR T cell expansion with response69 and contribution of T cell phenotypic subgroups with capacity to proliferate and persist long term70. Additionally, important insights into the roles of IL-6 and IL-1 in cytokine release syndrome and neurotoxicity71,72 and the contribution of a pan-T cell infiltrate and high cytokine levels in the CNS as mediators of neurotoxicity 73, have been gained by our group and others. However, there is a significant unmet need to apply a systematic approach interrogating the determinants of a successful response, toxicity, interaction with the endogenous immune system and short- and long-term effects of interventions aimed at reducing toxicity such as administration of the IL6R-antagonist Tocilizumab or IL-1 blockade74.

In this study we aim to systematically interrogate the characteristics of cell therapy products, evolution after administration in vivo and behavior in different compartments such as peripheral blood, bone marrow, CNS and if applicable tissues and their interplay with the endogenous immune system. Single cell transcriptomics, coupled with TCR-sequencing (when applicable BCR sequencing) and phenotypic characterization of transferred and endogenous immune cells as well as analysis of secreted immune factors such as cytokines, chemokines and antibodies in the plasma will be employed and correlated with clinical responses. This unbiased, systematic precision-diagnostic approach will allow identification of critical pathways which are common or distinct depending on the nature of the cell therapeutic approach, target and disease entities and associated or segregable from undesired toxicities. This will critically inform future rational design of cellular therapeutics and inform possible therapeutic interventions after cell therapy administration.

Vaccine Responses: A common theme among stem cell and solid organ transplant recipients, patients with current or prior malignancy, and patients with autoimmune or rheumatologic disease, including IBD, is impaired immune regulation, which is often compounded by the effect of immune-modifying treatments, including radiation, chemotherapy, and long-term immunosuppression. 15% of solid organ transplant recipients are hospitalized with a vaccine-preventable illness in the first five years after transplant in spite of measures to immunize these patients (Feldman et al., 2019), which is consistent with studies showing impaired responses to vaccines in these patients (Madan et al., 2008; Mazzone et al., 2004). HCT recipients respond to variable degrees to vaccination, but do not mount the same magnitude of response as in healthy controls, and may have further altered responses if they also have GVHD (Avetisyan et al., 2008; Shalabi et al., 2019). Patients with rheumatologic or autoimmune disease have also been shown to have impaired responses to particular vaccines, especially if on immunomodulatory agents such as TNFalpha blockade (Dell' Era et al., 2011). Studies of childhood cancer survivors suggest that immune impairment may persist beyond disease resolution; pediatric leukemia survivors who do not receive HCT have impaired humoral and adaptive immunity at treatment completion(Perkins et al., 2017; Top et al., 2020), and some patients do not respond, and others may have waning immunity(Nilsson et al., 2002; Top et al., 2020) in spite of re-vaccination attempts. As immunization efforts against SARS-CoV-2 become widespread, insight on the vaccine response in immunocompromised patients will be critical to informing more effective strategies to protect this population from severe COVID-19, which can be extrapolated to other vaccine-preventable pathogens.

In this study we propose to use a systematic approach to longitudinally profile humoral and antigen-specific T and B cell responses following SARS-CoV-2 vaccination in patients with a broad range of immune-modifying diseases. Blood samples from patients will be collected prior to, and at regular intervals following, vaccination. We will assess the durability and magnitude of long-term antibody responses using isotype-specific ELISAs and neutralizing antibody assays. High-parameter flow cytometry and scRNAseq will enable high-resolution phenotyping of antigen-specific T and B cell memory cells, as well as repertoire analysis, which may impact the likelihood of immune escape in vaccinated patients. Finally, this study will allow us to determine whether cloned antibodies or serum from patients with immune dysregulation are less able to neutralize viral variants, providing insight on whether reduced clonal diversity in patients may result in less protection against viral variants.

ELIGIBILITY:
A. Inclusion criteria for HCT patients:

1. Patients must be at least 1 month old and weigh >/= 3 kg.
2. Patients receiving any allogeneic or autologous hematopoietic stem cell transplantation (bone marrow, peripheral blood, or cord blood transplant).
3. Patients and/or parents or legal guardians must sign a written informed consent.

B. Inclusion Criteria for Adoptive Cellular Therapy (CT) patients:

1. Weight ≥3 kg
2. Patients receiving adoptive cellular therapy
3. Patient and/or legal guardian must sign written informed consent

C. Inclusion criteria for Healthy Donor Blood volunteers:

1. Age 18+
2. Participant does not have signs/symptoms of present illness
3. Participant does not have a known disease affecting the immune system
4. Participant is not on any medication/s that suppress immune system
5. Obtain informed consent

D. Inclusion criteria for HCT Related and Unrelated Donors:

1. Age >1 years of age
2. Weight >3 kg
3. Obtain informed consent

E. Inclusion criteria for IBD & FGID patients:

1. Patients must be at least 6 years old and weigh >/= 10 kg.
2. Patients being evaluated for IBD (new diagnosis or follow up of established disease), OR
3. Patients being evaluated for FGID (new diagnosis or follow up of established disease).
4. Obtain informed consent

F. Inclusion criteria for HCT & Cell Therapy Household Members:

1. Household member of a patient who is receiving HCT or Cell Therapy and who is participating in the PREDICT study
2. Age >1 years of age
3. Weight >3 kg
4. Obtain informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HCT, Cellular Therapy and Non-HCT patients undergoing endoscopy (patients with IBD and FGID) will be recruited from participating centers. This prospective banking study will continue to enroll patients undergoing HCT, endoscopy for IBD or FGID, and cellular therapy on an ongoing, long-term basis. Additional enrollment will come from patients receiving SARS-CoV-2 vaccination after HCT, solid organ transplant, active or recent malignancy or autoimmune or rheumatologic diagnoses, including patients who did not meet eligibility criteria for other cohorts. Additional patients who are healthy blood or bone marrow donors and may or may not be related to the patients with immune dysfunction or receiving HCT will also be enrolled in the study to serve as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Perform flow cytometry, TCR deep sequencing and whole transcriptome analysis on T cells purified from GI endoscopy samples taken for presumed GI GVHD, inflammatory bowel disease (IBD), and functional gastrointestinal disease (FGID). | 1 year
  To identify the mechanisms specific for auto-immune and allo-immune GI disorders.
Perform flow cytometry, TCR deep sequencing and transcriptome analysis on T cells from the peripheral blood in patients diagnosed with GI GVHD, IBD and FGID and patients receiving cellular therapies. | 1 year
  To identify the mechanisms specific for allo- and auto-immune diseases and the consequences of cellular therapy delivery.

SECONDARY OUTCOMES:
Perform longitudinal immune analysis on T cells and B cells purified from patients with allo- and auto-immune diseases and those receiving cellular immunotherapies. | 1 year
  Characterize the immunologic dysregulation responsible for auto- and allo-immune diseases and cellular therapies.
Perform microbiome analysis longitudinally in patients with auto- and allo-immune diseases. | 1 year
  Characterize the immunologic dysregulation responsible for auto- and allo-immune diseases.
Perform longitudinal immune analysis on T- and B-cells as well as measurements of serum antibody titers from patients with allo- and auto-immune disorders who receive immunization against COVID-19. | 1 year
  To identify immunologic determinants of response to COVID-19 immunization in patients receiving immunosuppressive therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Kean, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified Genomic data and clinical outcomes will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available in approximately 3 years and will be available thereafter for a period of 10 years.
Access Criteria: CITI and other ethics training, data transfer agreement with study sponsor.

REFERENCES:
- [Derived] Kaminski J, Fleming RA, Alvarez-Calderon F, Winschel MB, McGuckin C, Ho EE, Eng F, Rui X, Keskula P, Cagnin L, Charles J, Zavistaski J, Margossian SP, Kapadia MA, Rottman JB, Lane J, Baumeister SHC, Tkachev V, Shalek AK, Kean LS, Gerdemann U. B-cell-directed CAR T-cell therapy activates CD8+ cytotoxic CARneg bystander T cells in patients and nonhuman primates. Blood. 2024 Jul 4;144(1):46-60. doi: 10.1182/blood.2023022717. PMID 38558106